CLINICAL TRIAL: NCT01564654
Title: A Retrospective, Multi-Center Study to Evaluate the ConforMIS iTotal® CR (Cruciate Retaining) Total Knee Replacement System
Brief Title: A Retrospective Study of the iTotal CR Knee Replacement System
Status: Completed | Type: Observational
Sponsor: Restor3D (Industry)
Responsible Party: Sponsor
Other Study IDs: CCP 11-002
Record Dates: First submitted 2012-03-26; First posted 2012-03-28 (Estimated); Results first posted 2021-01-20 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- iTotal KRS
  Interventions: Device: iTotal KRS

INTERVENTIONS:
Device: iTotal KRS — Total Knee Replacement System

SUMMARY:
This study involves retrospective collection of data regarding the first approximately 100 iTotal Knee Replacement System surgeries and their short term outcomes at a small set of centers throughout the US.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical condition included in the approved Indications For Use
2. Has signed the informed consent form to allow review of medical records and collection of data therein.
3. > 18 years of age

Exclusion Criteria:

1. Treatment with iTotal in a manner inconsistent with Instructions for Use
2. Unwilling to sign then informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have received an iTotal Knee replacement
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - STAR Orthopedics, La Quinta, California
  - Preferred Orthopedics of the Palm Beaches, Boynton Beach, Florida
  - Tennessee Orthopaedic Alliance, Nashville, Tennessee
  - Central Utah Clinic, Provo, Utah

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | iTotal KRS
Started | 89 (106 knees (bilateral))
Completed | 89 (106 knees (bilateral))
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 106 knees (bilateral)
Arm/Group | iTotal KRS
Number analyzed (Participants) | 89
Age, Customized [Mean (Full Range); unit: years]
  Mean age at surgery | 68 [42 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 36

OUTCOME MEASURES:

1. Primary Outcome: Knee Function
Description: Range of Motion
Time Frame: Average of 7 months post-operative
Measure: Mean (Full Range); unit: degrees
Units Other Than Participants: Knees
Arm/Group | iTotal KRS
Number analyzed (Participants) | 89
Number analyzed (Knees) | 106
degrees | 113 [65 to 140]

2. Secondary Outcome: Revision Rate
Description: Number of knees that required a reoperation to remove/replace/add implant components
Time Frame: Average of 7 months
Population: bilaterals were included
Measure: Count of Units; unit: Knees
Units Other Than Participants: Knees
Arm/Group | iTotal KRS
Number analyzed (Participants) | 89
Number analyzed (Knees) | 106
Knees | 1

3. Secondary Outcome: Number of Transfusions
Description: Number of knees that required a blood transfusion during the initial hospital stay post-operative
Time Frame: Initial hospital stay
Measure: Number; unit: number of knees requiring transfusion
Units Other Than Participants: Knees
Arm/Group | iTotal KRS
Number analyzed (Participants) | 89
Number analyzed (Knees) | 106
number of knees requiring transfusion | 0

4. Secondary Outcome: Manipulations Under Anesthesia
Description: Number of knees that required a subsequent procedure to restore knee range of motion
Time Frame: Up to 7 months post-operative
Measure: Count of Units; unit: Knees
Units Other Than Participants: Knees
Arm/Group | iTotal KRS
Number analyzed (Participants) | 89
Number analyzed (Knees) | 106
Knees | 4

ADVERSE EVENTS:
Arm/Group | iTotal KRS
Serious Adverse Events (participants affected / at risk) | 5/89
Other Adverse Events (participants affected / at risk) | 0/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | iTotal KRS (N=89)
Manipulations (Surgical and medical procedures) | 4 (4)
Revision/Poly Swap (Surgical and medical procedures) | 1 (1) — Thicker insert implanted at 11 months post-op

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days